CLINICAL TRIAL: NCT04577521
Title: Prospective Single Centre Open Label Investigator Initiated Clinical Study to Evaluate the Efficacy and Safety of Cross-linked Intra-Articular Hyaluronic Acid (HA)(Biovisc Ortho Single) in Patients With Knee Osteoarthritis (OA)
Brief Title: The Safety and Efficacy of Single IA-HA Injection in Patients With Knee Osteoarthritis: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Goztepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Esat UYGUR, Assoc. Prof. MD, Goztepe Training and Research Hospital
Other Study IDs: 001
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BioVisc Ortho Single — BioVisc Ortho Single consisted of a prefilled syringe containing 90 mg/3 mL of IA-HA and is an injectable-grade HA from a biofermentation origin. Biovisc ortho single prefilled syringes are intended for single-use only, and the entire content of the syringe was injected into the target joint.

SUMMARY:
This prospective study was planned to carried out among the patients with grade II and III (Kellgren Lawrence classification) osteoarthritis of the knee attending outpatients clinic to evaluate the effectiveness and safety of viscosupplementation with intra-articular hyaluronic acid injection.

DETAILED DESCRIPTION:
The study was designed as prospective, single-center, single-arm, open-label, observational study. The patients with grade II and III (Kellgren Lawrence classification) osteoarthritis of the knee attending outpatients were planned to enroll the study. Patients between the age 18-80 years who did not achieve remission of pain despite receiving the first-line treatment for gonarthrosis including nonsteroidal anti-inflammatory drugs medication, activity modification and ice, were planned to included in the study. A single dose of HA will be injected into the target knee joint. Clinical evaluation will be done using the Western Ontario and McMaster Universities Arthritis Index (WOMAC) and the short form-36 questionnaires (SF-36 v2) at baseline, 3 months and 6 months by a clinical secretariat.

ELIGIBILITY:
Inclusion Criteria:

* Patients Age should not be less than 18 years.
* Patients must be able to understand and follow the study procedures and must provide written informed consent.
* Radiologically Grade II or III osteoarthritis of knee according to the Kellgren and Lawrence classification.
* Mild to moderate documented diagnosis of knee osteoarthritis that fulfill the ACR (American College of Rheumatology) criteria.
* Patients with consistent symptoms (joint pain, crepitus, swelling, effusion alone or combination of these symptoms) of knee osteoarthritis for at least 3 months prior to screening. If bilateral knee pain is present, the more painful knee will be selected.
* Patients who are willing to discontinue all non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesic medication taken for any condition, including their knee pain. However patients will be allowed to use only acetaminophen or aspirin as a rescue pain medication during the study period. The patients must abstain from medication use 24 hours prior to any study visit.

Exclusion Criteria:

* Patients with secondary osteoarthritis of the knee according to ACR criteria.
* Pregnant or lactating women, and women of childbearing potential not willing to use adequate contraception.
* Patients unable to stay in the study for 6 months, non- cooperating, not able to understand
* Patients having previously undergone surgery on target knee, including arthroscopy.
* Patients with neurological deficit in the lower extremities, with primary inflammatory joint disease, intra-articular tumours.
* Any severe systemic disease(s).
* Any significant osteoarthritis symptoms in other joints apart from the target knee which may require pharmacological treatment during the study.
* Patients who have received intra-articular hyaluronic acid within the previous 6 month and/or intra-articular steroids or articular lavage in the target knee within the previous 3 months prior to their inclusion in the study.
* Administration of glucosamine sulphate, chondroitin sulphate and diacerein within the 3 months prior to their inclusion in the study.
* History of allergy or hypersensitivity to hyaluronic acid.
* Participation in any clinical study in the last 3 months and any surgery scheduled in the next 8 months that can affect directly the result of the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with grade II and III (Kellgren Lawrence classification) osteoarthritis of the knee attending outpatients clinic
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 3 Months and 6 Months in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 3 Months and 6 Months
  WOMAC is health status measure questionnaire of twenty-four questions comprising 3 subscales (pain, stiffness and physical function). WOMAC was measured on a scale of 0-100 mm, where lower score represents lower pain and higher score represents higher pain.
Overview of Adverse Events (AE) | Through study completion, an average of 6 Months
  An AE could be any unfavorable and unintended symptom, sign, disease or condition, or test abnormality whether or not considered related to the investigational product. A serious adverse event (SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAE): AEs that developed/worsened during the 'on treatment period' (from first dose of study device until the end of study period). Category "AE" included participant with both serious and non-serious AE.

SECONDARY OUTCOMES:
Change in quality of life measured by SF-36 questionnaire (Short Form Health Survey questionnaire) | Baseline,3 Months and 6 Months
  36-Item Short Form Health Survey (SF-36) is a set of generic, coherent, and easily administered quality-of-life measures.each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided